CLINICAL TRIAL: NCT02006134
Title: Chronic Childhood Vasculitis: Characterizing the Individual Rare Diseases to Improve Patient Outcomes
Brief Title: Pediatric Vasculitis Initiative
Acronym: PedVas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: BC Childrens Hospital Research Institute (Unknown); University of Oxford (Other)
Responsible Party: Principal Investigator, David Cabral, Principle Investigator, University of British Columbia
Other Study IDs: H12-00894; TR2-119188 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-11-27; First posted 2013-12-10 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Wegeners Granulomatosis (Granulomatosis With Polyangiitis); Microscopic Polyangiitis; Eosinophilic Granulomatosis With Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis; Primary CNS Vasculitis; Unclassified Vasculitis
Keywords: Vasculitis; Primary CNS Vasculitis; Systemic vasculitis; Churg-Strauss Syndrome; Polyarteritis Nodosa; Wegener Granulomatosis; Pediatric vasculitis; Childhood vasculitis; Granulomatosis with polyangiitis; Microscopic Polyangiitis; Takayasu Arteritis; Autoimmune; ANCA-associated vasculitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa; Takayasu Arteritis; Vasculitis, Central Nervous System; Vasculitis; Systemic Vasculitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, biopsy tissue, urine, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PEDIATRIC VASCULITIS/PROSPECTIVE: Pediatric patients in this cohort are those diagnosed with vasculitis within 12 months from study entry. Clinical data, blood (RNA, plasma, serum), urine, and saliva (DNA) will be collected at 3 to 5 timepoints: time-of-diagnosis, post-induction, 12-month post diagnosis, disease flare, and remission/post-flare.
- PEDIATRIC VASCULITIS/RETROSPECTIVE: Patients in this cohort are those diagnosed with vasculitis more than 12 months from study entry and/or were previously enrolled in the ARChiVe or Brainworks registries. Clinical outcome data will be collected retrospectively. Blood (RNA & serum), urine, and saliva (DNA) will be collected at 2 timepoints: disease flare, and remission/post-flare.

SUMMARY:
Childhood chronic vasculitis describes a group of rare life-threatening diseases that have in common inflammation of blood vessels in vital organs such as kidneys, lungs and brain. Most knowledge about them comes from adult patients. Severe disease requires aggressive life-saving treatments with steroids and some cancer drugs which can themselves cause damage, and increase risks of cancer and severe infections. Conversely, milder disease can be treated with less toxic drugs. Different classification and "scoring tools" are used to define the types and severity of vasculitis and to measure damage caused by disease or drugs. These in turn help direct how aggressively to treat a patient and to measure outcome. None of these tools however have been assessed in children and the best balance of disease and treatment risks against outcome for children is not known. Although causes of these diseases in children and adults are probably the same, the effects of the disease and the response (good and bad) to drugs will differ in growing children. Because specialists may see only one new child with vasculitis each year, obtaining enough information to learn about childhood vasculitis requires cooperation. We will use an international web-based registry to which doctors from 50 or more centers can contribute patient data. We will determine the features which help better classify and diagnose children compared to adults. Through the web we will collect and analyze information on patients similarly classified and "scored" so that most successful treatments can be identified. Children with vasculitis are less likely to have diseases associated with aging, alcohol and smoking etc., and therefore may be a better group in whom to study the underlying biology of vasculitis. We will use this opportunity and collect spit, blood and tissue from registry patients for laboratory study with an aim to find biomarkers to better classify, define and direct optimal treatment and outcomes.

DETAILED DESCRIPTION:
We anticipate enrollment and collection of clinical data from as many as 600 children with various forms of childhood vasculitis, with approximately one third (200) of those children also contributing biological samples for study.

For children with vasculitis who are enrolled in the study, clinical information will be obtained from the medical chart from the time of diagnosis, post-induction (3-6 months post diagnosis) visit, 12-month clinic visit, and their most recent clinic visit or last clinic visit before discharge to adult care (ie. final outcome visit). Information that will be collected includes laboratory test results, biopsy and imaging results, disease activity, clinical history, and medications. Blood, urine, and saliva samples will also be collected at each clinic visit. If the subject experiences a disease flare, clinical data and biological samples will be collected at the time of the flare and at a later date when the disease remits.

The PedVas study is linked to an adult vasculitis initiative called DCVAS: Diagnosis and Classification Criteria in Vasculitis. Our DCVAS co-investigators and collaborators will recruit up to 250 adults at or near the time of diagnosis of the following forms of vasculitis: GPA, MPA, EGPA, TA, and UCV. Clinical data will be collected as part of the DCVAS study; this includes information such as laboratory test results, disease activity, and clinical history. Blood will also be collected and analyzed in parallel with samples collected from children with vasculitis. Finally, a DNA-biobank will be created and will house samples from approximately 700 adults and representing all forms of vasculitis. Recruitment will proceed according to DCVAS approved protocols and it will be conducted at participating DCVAS centres after the patient has formally consented to participation in the DCVAS study.

All biological samples will be processed and analyzed in Vancouver at the BC Children's Hospital Research Institute and at the University of British Columbia. Detailed data will be collected in electronic format and include demographic variables, socioeconomic status, detailed clinical history & physical findings, anthropometric measures, and measures of disease activity. All data for systemic vasculitis patients will be directly entered at each site into a secure, online, web-based data entry system called REDCap which is managed through the data management centre at the University of British Columbia in Vancouver.

ELIGIBILITY:
Inclusion criteria for vasculitis subjects:

* Diagnosed with ANCA-associated vasculitis (AAV: such as Granulomatosis with Polyangiitis (GPA), Eosinophilic Granulomatosis with Polyangiitis (EGPA) and Microscopic Polyangiitis (MPA)), Primary Angiitis of the Central Nervous System (PACNS), Unclassified vasculitis, Takayasu's Arteritis (TA) or Polyarteritis Nodosa (PAN) before age 18

Inclusion criteria for healthy controls:

* Healthy adult or child

Exclusion Criteria for vasculitis subjects:

* Diagnosed with other vasculitis subtypes not listed above
* More than 20 years of age

Exclusion criteria for healthy controls:

* Donated greater than 20 ml of blood in the previous three weeks
* Has an immune disorder or blood borne infectious diseases (such as HIV or Hepatitis)
* Has vasculitis, multiple sclerosis, diabetes, an autoimmune disease, a thyroid condition, or other chronic conditions involving the heart, lungs, gut or kidney
* Has a previous history of anaemia or abnormal blood clotting
* Has a current or previous drug abuse problem

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children or adolescents diagnosed with vasculitis at any of the participating PedVas study centres
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2013-01; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Develop new benchmarks for outcome in pediatric patients with systemic vasculitis | within 3 yrs
  Specific and generic disease assessment tools will be used to analyze our registry cohorts to enable the first-ever benchmarks of outcome in children with GPA who have had a minimum of 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: David Cabral, MBBS, Principal Investigator — University of British Columbia; BC Children's Hospital; Raashid Luqmani, DM FRCP(E), Principal Investigator — University of Oxford; Dirk Foell, MD, Principal Investigator — Universität Münster; Robert Hancock, PhD, Principal Investigator — University of British Columbia; Colin Ross, PhD, Principal Investigator — University of British Columbia
Locations (32):
- United States (10):
  - University of San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Comer Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - The Joseph M. Sanzari Children's Hospital, Hackensack, New Jersey
  - Children's Hospital at Montefiore, The Bronx, New York
  - Akron Children's Hospital, Akron, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Utah / Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (8):
  - University of Calgary / Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Janeway Childrens Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IIWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Rigshospitalet, Copenhagen, Denmark
- University Children's Hospital, Münster, Germany
- Sanjay Gandhi Post Graduate Institute, Lucknow, India
- Siriraj Hospital, Bangkok, Thailand
- United Kingdom (10):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Royal Hospital for Children, Glasgow
  - Leeds Children's Hospital, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne
  - Nottingham Children's Hospital, Nottingham
  - Nuffield Orthopaedic Centre, Oxford
  - Sheffield Children's Foundation Trust, Sheffield
  - Southampton General Hospital, Southampton

REFERENCES:
- See also: BrainWorks: The International Childhood CNS Vasculitis Outcome Study — http://www.sickkids.ca/Research/Brainworks/the-brainworks-study/index.html
- See also: DCVAS: Diagnostic and Classification Criteria in Vasculitis Study — https://research.ndorms.ox.ac.uk/public/dcvas/